CLINICAL TRIAL: NCT06015789
Title: Self-care in Patients Affected by Inflammatory Bowel Disease and Caregivers' Contribution to Self-care
Acronym: IBD-Self
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5886 - IBD-Self
Record Dates: First submitted 2023-08-02; First posted 2023-08-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Administration of questionnaires for the evaluation of self-care

SUMMARY:
The Inflammatory Bowel Disease (IBD) is a chronic inflammatory disease of the gastrointestinal tract including Crohn's disease and Ulcerative Colitis. The course of IBD is frequently progressive and can be hardly predictable, with sudden exacerbations of intestinal symptoms. Epidemiological studies have shown that IBD has an increasing prevalence to reach 10 million people in 2030. These diseases require frequent interactions between patients and the healthcare system, or symptom management with continuous therapies, gastroenterological visits, surgery, contacts for resolution of urgent symptoms from telephone and email, access to the emergency, hospitalizations, nutritional counseling, psychological interventions and follow-up controls. An IBD can completely disrupt a family's ability to function normally and often imposes a strain on family members' relationships. In the model of self-care in chronic diseases, according to Riegel's "Middle Range Theory", there are external factors, predictive factors that can influence and limit the patient's attitude and therefore his self-esteem, the ability to implement decision-making behaviors to improve and increase his self-care. There are also factors that influence a person's self-care decisions: the particular caregivers. In this process, the role of the caregiver and the dyad he establishes with the patient can influence the whole process of self-confidence and self-care. The objectives of the study are to investigate and describe self-care in patients with IBD and how their caregivers in dyadic interaction can contribute.

DETAILED DESCRIPTION:
Study design Multicentre prospective observational study

Population The study is multicentre and will be conducted at the Fondazione Policlinico Gemelli IRCCS in Rome as the reference centre together with the centres that decide to participate. Patients will be enrolled at the IBD centres, in the medical wards, during visits or during hospitalization. Follow-up will be after the first administration at T1 (6 months) and T2 (12 months). Subsequent questionnaires (T1 and T2) will be administered by telephone or telematically. The study will start as soon as it is approved by the Ethics Committee. The total duration of the study will not exceed 12 months from the last enrolment.

Duration of the study The study will last 12 months from the date of approval by the Ethics Committee. The study is hypothetically expected to be completed by the end of December 2024.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older;
* voluntary participation in the study;
* patient with the diagnosis of IBD outpatients and non-hospitalized;
* caregiver of patients with IBD diagnosis outpatients and hospitalised;
* Reading and signing informed consent

Exclusion Criteria:

* patients with a diagnosis of IBD for less than 12 months;
* caregivers of patients with an IBD diagnosis for fewer than 12 months;
* patients operated for less than 6 months; care providers of patients operating less than six months;
* reduced mastery of the Italian language;
* subjects suffering from serious psychiatric disorders;
* serious clinical conditions that would not allow the completion of the questionnaire;
* refusal to sign the informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research is multicenter and will be conducted in the IBD units and in the medical departments of the centers that will decide to join, during visits or hospitalization. Male or female patient, adult.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the factors that affect the self-care of the patient with IBD, of the caregiver and of their dyadic interaction; | Day 0, 6 months, 12 months
  Evaluate through the administration of validated questionnaires the level of self-care of outpatient or inpatient IBD patients and their caregivers and correlate it with quality of life, anxiety, stress and other predictive factors

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Napolitano, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Daniele Napolitano, Rome, Italy

REFERENCES:
- [Derived] Napolitano D, Biagioli V, Bartoli D, Cilluffo S, Martella P, Monaci A, Vellone E, Cocchieri A. Validity and Reliability of the Self-Care of Chronic Illness Inventory in Patients Living With Inflammatory Bowel Disease. J Clin Nurs. 2025 Nov;34(11):4642-4653. doi: 10.1111/jocn.17712. Epub 2025 Mar 3. PMID 40033448
- [Derived] Napolitano D, Vellone E, Iovino P, Scaldaferri F, Cocchieri A. Self-care in patients affected by inflammatory bowel disease and caregiver contribution to self-care (IBD-SELF): a protocol for a longitudinal observational study. BMJ Open Gastroenterol. 2024 Aug 29;11(1):e001510. doi: 10.1136/bmjgast-2024-001510. PMID 39209770